CLINICAL TRIAL: NCT06662513
Title: An Australian Regional Hospital's Oesophagectomy Outcomes
Brief Title: Post Oesophagectomy Outcomes in a Single Regional Centre in Australia
Status: Not yet recruiting | Type: Observational
Sponsor: Launceston General Hospital (Other)
Collaborators: Department of Health, Tasmania (Other Government)
Responsible Party: Principal Investigator, Renishka Sellayah, Principal investigator, Launceston General Hospital
Other Study IDs: 2024/ETH01712
Record Dates: First submitted 2024-10-21; First posted 2024-10-29 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Oesophageal Cancer
Keywords: oesophageal cancer; regional surgery
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- oesophagectomy: patients who underwent oesophagectomy within the specified time frame
  Interventions: Other: No Intervention: Observational Cohort

INTERVENTIONS:
Other: No Intervention: Observational Cohort — No intervention - retrospective observational study

SUMMARY:
Literature review/rationale for project

* Oesophageal cancer is associated with a grim prognosis despite many advances in treatment. Oesophagectomy is a key component of the care of patients who are candidates for curative treatment, however it is associated with substantial morbidity.
* Several studies have suggested that oesophagectomies performed at higher volume tertiary centres are associated with lower morbidity and mortality than lower volume centres, and this has prompted changes to policy in countries such as Great Britain, Canada and the Netherlands with regards to the centralisation of these cases. A higher volume centre within Australia is likely to perform 6 or more procedures per year.
* Currently within Australia, centralisation on a large scale has not occurred. This has been limited in part by resource provision and geographical barriers. Therefore, oesophagectomies in Australia are still routinely performed in regional centres. However, there is a paucity of recent outcomes data from these centres.

Aims/objectives

* Retrospective review of oesophagectomies undertaken in a single regional centre in Tasmania, Australia over 10 years (January 2014 to December 2023)
* Assess outcomes (long and short-term complications and mortality) and compare to morbidity and mortality rates from larger international centres

DETAILED DESCRIPTION:
Research aims/objectives

* Retrospective review of oesophagectomies undertaken in a single regional centre in Tasmania, Australia over 10 years (January 2014 to December 2023)
* Assess outcomes (long and short-term complications, mortality, survival) and compare to published outcomes from larger national and international centres

Project Design Research project setting: Launceston General Hospital (Tasmania, Australia)

Methodological approach: Retrospective case series

Participants

* Retrospective identification of patients who underwent oesophagectomy at Launceston General Hospital from January 2014 to December 2023 via coding in medical records and MBS codes
* Inclusion criteria: patients who underwent oeosphagectomy at LGH in the specified time frame
* Exclusion criteria: none
* Expected size of case series is approximately 100 patients (this is extrapolated from the number of oesophagectomies performed in 2023)

Participant recruitment strategies and timeframes: No active participation of patients in this case series, all information will be retrospectively collected from medical records

Consent: Given the number of expected patients (approximately 100) and the potential distress that could be caused to patients or their next of kin in seeking consent, an Application for the Waiver of the requirement for Consent will be submitted

Research Activities

* No participant commitment is required
* Project duration is approximately 4 weeks for data collection, 4 weeks for analysis and writing
* No Participant follow-up is planned as part of this project

Data Collection/Gathering

* Data will be collected by assessment medical records only
* Only the PI will access identifying details such as name and date of birth.
* Information that will be collected includes: Patient demographics: age, gender, neoadjuvant treatment, co-morbidities, BMI, ASA score, type of oesophagectomy (2 or 3 stage). Primary endpoints: mortality (in hospital, 30 day and 90 day), anastomotic leak, length of stay (ICU, acute inpatient). Secondary endpoints: chyle leak, pneumonia, reintubation, return to theatre, wound infection, intra-abdominal infection, cardiac complications, DVT/PE, anastomotic stricture, diaphragmatic hernia, disease recurrence, survival

Data Management

* Data will be entered into an excel spreadsheet kept on a password protected THS computer in the department of surgery in LGH
* Data will only be accessed by the named investigators that are based at LGH (no external researcher will have access to data)
* There will be no hard copies of this data
* Data will not be transferred to personal computers/laptops
* Data will be destroyed/deleted by the PI 5 years after publication date

Data Analysis

* Outcomes will be calculated as percentages and then compared to published outcomes data from other Australian centres and international centres Examples of some published studies that may be used to compare outcomes are listed in citations.
* Given the retrospective nature of the data collection it is anticipated that some information will be missing however the kind of data the investigators plan to collect is very likely to be found in the medical record.
* Any missing information will be acknowledged when assessing results and the impact of the missing information will also be acknowledged when making any conclusions from those results

ELIGIBILITY:
Inclusion Criteria:

* patients who underwent oeophagectomy at Launceston General Hospital between January 2014 to December 2023

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients who underwent oeophagectomy at Launceston General Hospital between January 2014 to December 2023
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2024-11-14 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
mortality | from date of surgery to end of study (November 2024) for a timeframe up to 10 years
  date of death from any cause or date of palliation whichever came first
Anastomotic leak | from date of surgery to end of study period (Nov 2024), assessed up to 10 years
  Grade 1-3, diagnosed radiologicaly, requiring intervention (surgical or non-surgical)
Length of stay | from date of surgery to discharge date of hospital admission, approximately 2-4 weeks in most cases but assessed up to 12 weeks
  total inpatient hospital stay and total ICU length stay

CONTACTS AND LOCATIONS:
Locations (1):
- Launceston General Hospital, Launceston, Tasmania, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chang AC. Centralizing Esophagectomy to Improve Outcomes and Enhance Clinical Research: Invited Expert Review. Ann Thorac Surg. 2018 Sep;106(3):916-923. doi: 10.1016/j.athoracsur.2018.04.004. Epub 2018 May 5. PMID 29738757
- [Background] Pu S, Chen H, Zhou C, Yu S, Liao X, Zhu L, He J, Wang B. Major Postoperative Complications in Esophageal Cancer After Minimally Invasive Esophagectomy Compared With Open Esophagectomy: An Updated Meta-analysis. J Surg Res. 2021 Jan;257:554-571. doi: 10.1016/j.jss.2020.08.011. Epub 2020 Sep 11. PMID 32927322
- [Background] De Silva I, Wee M, Cabalag CS, Fong R, Tran K, Wu M, Schloithe A, Bright T, Duong CP, Watson DI. Para-conduit diaphragmatic hernia following esophagectomy-the new price of minimally invasive surgery? Dis Esophagus. 2023 Apr 29;36(5):doad011. doi: 10.1093/dote/doad011. PMID 36912068
- [Background] Buchholz V, Hazard R, Lee DK, Liu DS, Zhang W, Chen S, Aly A, Barnett S, Le P, Weinberg L. Textbook outcomes after oesophagectomy: a single-centre observational study. BMC Surg. 2023 Dec 8;23(1):368. doi: 10.1186/s12893-023-02253-7. PMID 38066440
- [Background] Edmondson J, Hunter J, Bakis G, O'Connor A, Wood S, Qureshi AP. Understanding Post-Esophagectomy Complications and Their Management: The Early Complications. J Clin Med. 2023 Dec 11;12(24):7622. doi: 10.3390/jcm12247622. PMID 38137691
- [Background] Oesophago-Gastric Anastomosis Study Group on behalf of the West Midlands Research Collaborative. Comparison of short-term outcomes from the International Oesophago-Gastric Anastomosis Audit (OGAA), the Esophagectomy Complications Consensus Group (ECCG), and the Dutch Upper Gastrointestinal Cancer Audit (DUCA). BJS Open. 2021 May 7;5(3):zrab010. doi: 10.1093/bjsopen/zrab010. PMID 35179183
- [Background] Anderson O, Ni Z, Moller H, Coupland VH, Davies EA, Allum WH, Hanna GB. Hospital volume and survival in oesophagectomy and gastrectomy for cancer. Eur J Cancer. 2011 Nov;47(16):2408-14. doi: 10.1016/j.ejca.2011.07.001. Epub 2011 Aug 9. PMID 21835609
- [Background] Doran SLF, Digby MG, Green SV, Kelty CJ, Tamhankar AP. Risk factors for and treatment of anastomotic strictures after Ivor Lewis esophagectomy. Surg Endosc. 2024 Nov;38(11):6771-6777. doi: 10.1007/s00464-024-11150-w. Epub 2024 Aug 19. PMID 39160303